CLINICAL TRIAL: NCT05102500
Title: Examining the Decision-Making Process and Characteristics of Cancer Patients Who Sought Second Opinions at the University of Colorado
Brief Title: Second Opinions in Oncology
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 21-3100.cc
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Pancreatic Cancer; Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Chart Review Patients: The PI will conduct a retrospective chart review of breast cancer, colorectal cancer, and pancreatic cancer patients to better understand the patient, disease, and treatment characteristics that play a role in second opinion retention rates.
- Semi-structure Interview Patients: The PI will conduct semi-structured interviews with breast cancer, colorectal cancer and pancreatic cancer patients to better understand the decision-making process that goes into continued care with their primary or second opinion physician.

SUMMARY:
The long-time goal is to understand what decision-making process and patient characteristics factor into a patient deciding to stay with their initial physician versus seeking treatment with a second opinion.

DETAILED DESCRIPTION:
The long-time goal is to understand what decision-making process and patient characteristics factor into a patient deciding to stay with their initial physician versus seeking treatment with a second opinion. To do this, the PI will examine the second opinion retention rates and patient characteristics of three distinct populations: breast cancer patients, pancreatic cancer patients and colorectal cancer patients. The study team hypothesize the majority of breast cancer and colorectal cancer patients who seek a second opinion at the University of Colorado, will preferentially choose to return to their first provider, whereas patients with pancreatic cancer who seek a second opinion at the sponsor's institution will be more likely to go on to receive care at the University of Colorado. The PI predicts the difference in second opinion retention rates between these three populations is due to the ability of the second opinion pancreatic cancer provider's ability to offer more treatment or a different treatment plan at the sponsor institution relative to the patient's first provider. The study team also predict that socioeconomic status and education will have a positive correlation with changing to with a second opinion physician whereas geographic distance and treatment plan similarity will have a negative correlation. The study team will assess this hypothesis by conducting a retrospective cohort study of breast, pancreatic, and colorectal cancer patients who received a second opinion at the University of Colorado. From this cohort, the study team will identify patients who both received their care at the sponsor institution and patients who returned to their initial provider to receive care. The study team will invite these patients to participate in semi-structured interviews to better understand how and why the patient made their treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients who are 18 years of age or older who received a second opinion at the University of Colorado.
* A subset of these patients will be invited to participate in semi-structured interviews

Exclusion Criteria:

* Patients under the age of 18.
* Patients who did not receive a second opinion at the University of Colorado.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients who are 18 years of age or older who received a second opinion at the University of Colorado will be included in the retrospective chart review and analysis. A subset of these patients will be invited to participate in semi-structured interviews
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Second opinion retention rates for cancer patients at University of Colorado | 12 months
  a. The study team will perform a retrospective chart review to identify patients with breast cancer, colorectal cancer or pancreatic cancer who were seen by a surgeon at the University of Colorado for a second opinion and to examine whether or not the subject stayed at the Cancer Center to receive cancer care. The study team predict the second opinion retention rate - the percent of patients who received a second opinion at the Cancer Center and ultimately received care at this institution - will be significantly higher for pancreatic cancer patients than for breast and colorectal cancer patients.

SECONDARY OUTCOMES:
Univariate statistical analysis affecting second opinion retention rates | 12 months
  a. The study team will perform univariate analysis on patient, disease, and treatment characteristics for the second opinion patients who did and did not receive cancer care at this institution to identify factors associated with high and low second opinion retention rates. The study team hypothesize patient factors (socioeconomic status, education, and geographic distance), disease factors (more advanced disease or less common tumor subtypes), and treatment factors (offering more or different treatment) will affect the second opinion retention rates for breast and pancreatic cancer patients.

OTHER OUTCOMES:
Patient opinions on decision making process through semi-structure interviews | 12 months
  a. The study team will identify patients who both received their care at the second opinion institution and patients who returned to the initial provider to receive care. The study team will invite these patients to participate in semi-structured interviews to better understand how and why treatment decisions were made.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tevis, Principal Investigator — Colorado Research Center
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided